CLINICAL TRIAL: NCT05095740
Title: The Effects of Neuromodulation on Phonatory Function in Laryngeal Dystonia
Brief Title: Effects of Neuromodulation in Laryngeal Dystonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MGH Institute of Health Professions (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Teresa J Kimberley, Professor, MGH Institute of Health Professions
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020P003531; K24DC018603 (NIH)
Record Dates: First submitted 2021-02-15; First posted 2021-10-27 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Laryngeal Dystonia; Focal Dystonia
Keywords: transcranial magnetic stimulation; randomized control trial; rTMS
MeSH Terms: conditions — Dysphonia; Dystonic Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive 5 consecutive days of either rTMS or sham rTMS. Day 1, baseline (Pre) acoustic, perceptual and patient-reported assessments of voice production and TMS-measured neurophysiology will be performed. Participants will then receive the first rTMS intervention. Day 2, 3 and 4, participants will receive rTMS intervention solely, with no testing. Day 5, the same acoustic, perceptual, patient-reported and assessments will be performed after rTMS intervention. At least 3 months after Post1, participants will cross-over to receive the other intervention. Assessments in Pre2 and Post2, will mirror the timing of Pre1 and Post1 in phase 1. Following treatments, acoustic measures and a global rating of change in vocal function will be evaluated to understand the longevity of our treatment approach. Follow up voice recordings will be obtained using a portable voice recorder given to and returned by participants at their initial visit.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomly assigned to one of two arms of this study (real rTMS or sham). Only the study personnel tasked with setup of the rTMS equipment will know to which group each participant has been randomized so that they can adjust the machine parameters for each participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- repetitive transcranial magnetic stimulation (rTMS) (Active Comparator): 5 consecutive days of rTMS to the individualized, targeted, left laryngeal motor cortex associated with laryngeal function to down-regulate cortical motor signal to intrinsic laryngeal muscles and improve vocal function of individuals with LD.
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)
- Sham rTMS (Sham Comparator): 5 consecutive days of sham rTMS to the individualized, targeted, left laryngeal motor cortex associated with laryngeal function to down-regulate cortical motor signal to intrinsic laryngeal muscles and improve vocal function of individuals with LD.
  Interventions: Device: sham rTMS

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation (rTMS) — Repetitive transcranial magnetic stimulation used to regulate the contribution of the laryngeal motor cortex to voice production and laryngeal motor muscle activation.
  Other Names: transcranial magnetic stimulation
  Arms: repetitive transcranial magnetic stimulation (rTMS)
Device: sham rTMS — Repetitive transcranial magnetic stimulation used to a cortical area not associated with change in outcomes at an intensity substantially lower than that of the established threshold.
  Other Names: sham repetitive transcranial magnetic stimulation
  Arms: Sham rTMS

SUMMARY:
Laryngeal dystonia (LD) causes excessive vocal fold abduction (opening) or adduction (closing) leading to decreased voice quality, job prospects, self-worth and quality of life. Individuals with LD often experience episodic breathy voice, decreased ability to sustain vocal fold vibration, frequent pitch breaks and in some cases, vocal tremor. While neuroimaging investigations have uncovered both cortical organization and regional connectivity differences in structures in parietal, primary somatosensory and premotor cortices of those with LD, there remains a lack of understanding regarding how the brains of those with LD function to produce phonation and how these might differ from those without LD. Intervention options for people with LD are limited to general voice therapy techniques and Botulinum Toxin (Botox) injections to the posterior cricoarytenoid (PCA) and/or TA (thyroarytenoid) often bilaterally, to alleviate muscle spasms in the vocal folds. However, the effects of injections are short-lived, uncomfortable, and variable. To address this gap, the aim of this study is to investigate the effectiveness of repetitive transcranial magnetic stimulation (rTMS), a non-invasive neuromodulation technique, in assessing cortical excitability and inhibition of laryngeal musculature. Previous work conducted by the investigator has demonstrated decreased intracortical inhibition in those with adductor laryngeal dystonia (AdLD) compared to healthy controls. The investigators anticipate similar findings in individuals with with other forms of LD, where decreased cortical inhibition will likely be noted in the laryngeal motor cortex. Further, following low frequency (inhibitory) rTMS to the laryngeal motor brain area, it is anticipated that there will be a decrease in overactivation of the TA muscle. To test this hypothesis, a proof-of-concept, randomized study to down-regulate cortical motor signal to laryngeal muscles will be compared to those receiving an equal dose of sham rTMS. Previous research conducted by the investigator found that a single session of the proposed therapy produced positive phonatory changes in individuals with AdLD and justifies exploration in LD.

DETAILED DESCRIPTION:
The cause of LD is largely unknown and there are no treatments that produce long-term benefits. The investigators' long-term goal is to elucidate the pathophysiology of laryngeal dystonia as a crucial step towards the development of sensitive testing and novel interventions to treat this devastating disease. Neuroimaging studies have suggested that LD is associated with abnormal patterns of activation and excessive plasticity in sensorimotor areas in the brain, however, an understanding of the cortical excitability in this disorder is lacking. This information is important because it provides a more comprehensive understanding of the pathophysiology of the disorder, opening potential investigation into novel tests or treatments. The investigators have begun to address this gap in knowledge by developing a novel transcranial magnetic stimulation (TMS) paradigm to assess intracortical excitability and inhibition of targeted laryngeal muscles. Although similar paradigms have been fruitful for explicating the neural mechanisms of dystonia in the limbs, to our knowledge TMS has not been used to assess pathophysiology in laryngeal dystonia, thus similarities and differences in brain state between the limb and laryngeal dystonias could not be assessed. The investigators' current NIDCD project (R01DC015216) with which this proposed project synergizes, uses TMS and functional neuroimaging in people with LD and focal hand dystonia to determine the brain excitability and connectivity, distinctive of, and common to the two disorders. This approach is based on the investigators' recently completed NIDCD grant (R21DC012344) which supported the development of a valid and reliable TMS method to determine the cortical representation and excitability of the thyroarytenoid, a muscle affected in LD. Utilizing this approach, the investigators have recently demonstrated that people with LD have reduced intracortical inhibition compared to healthy controls. These results provide a compelling basis for the clinical application of this finding to determine if an intervention that increases intracortical inhibition can produce clinical improvements.

Aim 1: Determine the phonatory effects of 5-days of daily rTMS vs sham in people with LD. The effects of rTMS on phonatory function will be measured using (a) auditory-perceptual assessment (b) acoustic analysis including smoothed cepstral peak prominence (CPPS) of running speech and sustained vowel, and (c) patient self-ratings of vocal effort (response to voice demand). (H1) The investigators will observe large favorable intervention effect sizes in measures of phonatory function following rTMS compared to sham.

Aim 2: Determine the neurophysiologic changes associated with 5 days of rTMS vs sham in people with LD. The intervention effects on TMS-measured neurophysiology including intracortical excitatory and inhibitory measures from the laryngeal motor cortex will be assessed pre and post intervention. (H2) The investigators will observe significant decreases in cortical excitability [motor evoked potential (MEP)] and/or increases in inhibition [cortical silent period (cSP)] following rTMS compared to sham.

Aim 3: Explore characteristics associated with responders vs non-responders to rTMS in people with LD. This exploratory aim will stratify participants as responders or non-responders based on each person's acoustic (CPPS) changes. A multivariate regression will explore factors associated with positive response to intervention. (H3) Certain factors such as age, time since symptom onset, clinical severity, and/or baseline cortical excitability and inhibition will be associated with treatment responsiveness.

Procedures: Qualified participants will provide informed consent and receive on-site screening to determine eligibility. On Day 1, baseline (Pre) acoustic, perceptual and patient-reported assessments of voice production and TMS-measured neurophysiology will be performed. Participants will then receive the first rTMS intervention. On Day 2, 3 and 4, participants will receive rTMS (real or sham) intervention solely, with no testing. On Day 5, the same acoustic, perceptual, patient-reported and neurophysiologic assessments will be performed after rTMS intervention. At least 3 months after Post1, participants will cross-over to receive the other intervention (rTMS or Sham). The timing of the assessments in the cross-over phase of the experiment, Pre2 and Post2, will mirror the timing of Pre1 and Post1 in the first phase.

TMS Neurophysiology Assessment. Participants will have the vocalization area tested. Topical anesthesia will first be applied to the anterior neck skin followed by a superficial injection of 1% lidocaine with 1:100,000 epinephrine. The target muscles are bilateral TA muscles. A 30 mm, 27 gauge needle loaded with a pair of fine-wire hooked electrodes will be inserted into each TA muscle by an experienced otolaryngologist following standard procedures for laryngeal EMG. Using a percutaneous approach, the needle will be passed through the cricothyroid membrane at an angle off midline but medial to the ipsilateral inferior tubercle, to directly enter the TA muscle while avoiding the airway. During insertion, the electrodes are connected to an audio monitor to monitor muscle activity in real-time during placement. After the TA placement is confirmed, the needle is removed leaving the fine-wires in the TA muscles. The two pairs of fine-wire electrodes will be connected to the amplifier and acquired with the same setup that are reported in the investigators' previous study. electrode locations will be confirmed by increased EMG activity with sustained phonation and Valsalva maneuver. The TMS testing intensity threshold will be determined by finding the minimum intensity required to elicit a cortical silent period (cSP) during constant phonation of /i/ (to elicit contraction from the TA muscles) as a measure of cortical inhibition. The TMS 'hotspot' will be the corresponding location on the cortex when cSP is induced with the TMS testing intensity threshold. TMS hotspot location and 30 trials of fine-wire electrodes electromyogram (EMG) cSP response from TA muscle will be recorded. The cSP reflects GABAB receptor mediated inhibitory processes within cortical motor areas. Ten trials motor evoked potential (MEP) will also be evoked with the participants as rest as a measure of cortical excitability. EMG area under the curve will be calculated for a time-equivalent period of pre-stimulus activity. A frameless stereotactic neuro-navigation system will be used to enhance the reliability and recording of stimulus locations. To ensure safety, an investigator will screen each participant to determine appropriateness for TMS and that all safety parameters are met. Processing will occur according to previously published methods. The investigator performing the excitability assessment will be blind to group designation.

rTMS. Inhibitory (1 Hz) rTMS (1200 pulses, biphasic waveform) will be delivered to the same left hemisphere laryngeal motor cortical 'hotspot' established with the TMS testing on Day 1. The left laryngeal cortex was selected due to the bilateral nature of control of the laryngeal muscles, and findings of no difference between left and right sided cSP. Neuronavigation (Brainsight®, Rogue Research Inc. Quebec, Canada) will be used to enhance rigor by tracking stimulation location in the cortex and coil position as the stimulation target. Subject will receive approximately 20 minutes of FDA-approved rTMS treatment at 0.9 x resting motor threshold at 1 Hz with a 70-mm figure-eight TMS coil connected to 5Magstim rapid magnetic stimulator. This treatment is within the range for total pulses performed in previous studies in subjects with other dystonias in a single day. The same target will be used for the rTMS intervention over the 5 days and for the post-intervention assessments. Sham rTMS stimulation will be delivered with a sham coil that produces similar sound and sensory stimulation to the scalp but does not deliver a stimulating pulse. Sham stimulation will help deter mine whether the changes following rTMS are due to placebo effect.

ELIGIBILITY:
Inclusion Criteria:

* Age range is 21-85 years
* Diagnosis of Laryngeal Dystonia (LD)
* Subject is able to give informed consent
* Symptoms at worst severity if receiving botulinum toxin injections
* Subject has signed the consent form

Exclusion Criteria:

* Other forms of dystonia
* Vocal fold pathology or paralysis
* Essential tremor
* Laryngeal cancer or other neurologic conditions with medications affecting the central nervous system
* History of laryngeal surgery
* Adults lacking the ability to consent or complete the assessments and intervention
* Seizure in the last 2 years
* Contraindications to rTMS

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Objective Assessment of Phonatory Function | Day 1 (baseline), day 5 (post intervention), and Day 12 (follow up) timepoints for both arms of the study.
  Participants will produce sustained /ah/ vowels, read the rainbow passage and engage in freeform conversation. This speech will be recorded and measures of cepstral peak prominence smoothed (CPPS; range: 0-100, where higher indicates stronger voice signal and correlates highly with better voice quality).
Change in Cortical Excitability (intrahemispheric inhibition) | Day 1 (baseline), Day 5 (post intervention)
  Intrahemispheric inhibition will be measured with the cortical silent period (cSP) measured in ms

SECONDARY OUTCOMES:
Subjective Assessment of Phonatory Function | Day 1 (baseline), Day 5 (post intervention), and Day 12 (follow up) timepoints for both arms of the study.
  Three speech language pathologists who specialize in voice disorders and are blinded to treatment day or group, will listen to the recorded audio sentences and sustained vowels and perform an independent overall perceptual evaluation of each participant's voice for each assessment session using the rating scales from the American Speech-Language-Hearing Association recommended Consensus Auditory Perceptual Evaluation of Voice (CAPE-V). The primary measure will be the rating for Overall Severity of dysphonia, and secondary measures will include ratings for strain, roughness, breathiness, pitch and loudness. Scores closer to 0 indicate less severity and closer to 100 indicate more severely disordered. Each judge will listen to recordings of 20% of the assessments (randomly selected) twice for purposes of estimating intra-judge reliability. Ratings from the three judges will be averaged to produce one score for each perceptual parameter.
Self Ratings of Voice Effort | Day 1 (baseline), Day 5 (post intervention), and Day 12 (follow up) timepoints for both arms of the study.
  Self ratings of voice effort on a visual analog scale (VAS) after reading the sentences in Outcome 1. "Speaking required how much effort?" 0=minimal effort, 10= maximal effort
Secondary Objective assessment of phonatory function | Day 1 (baseline), Day 5 (post intervention), and Day 12 (follow up) timepoints for both arms of the study.
  In addition to the CPPS (primary measure above), the voice samples will be analyzed with the following: number of phonatory breaks (range: 0-x; were few breaks indicates a better voice quality), frequency shifts (range: 0-x Hz; where a smaller shift (closer to 0) is generally indicative of better voice quality) and the number of aperiodic segments (range: 0-x; where fewer aperiodic voice segments is generally indicative of better voice quality) will be obtained from each recording. These will be analyzed and compared over time.

OTHER OUTCOMES:
Forced choice paired assessment of phonatory function | Day 1 (baseline), Day 5 (post intervention), and Day 12 (follow up) timepoints for both arms of the study.
  If the primary or secondary assessments of objective or perceptual ratings of change fail to capture change in participants' voice between baseline and post intervention, a forced choice question will be posed to blinded raters to ask which paired voice sample represents the less severe sample and then perform a VAS ranking of how severe the voice sample sounds (0=minimal impairment, 10=severe impairment)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa J Kimberley, PhD,PT, Principal Investigator — MGH Institute of Health Professions
Locations (1):
- Teresa J Kimberley, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate technology; and (3) a commitment to destroying or returning the data after analyses are completed. Sharing and modification rights will be determined for individual users by the PI of this study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available no later than upon the acceptance of publication of the final dataset.
Access Criteria: Listed as personnel on Massachusetts General Hospital individualized health plan institutional review board for this study and as determined by the principal investigator.

REFERENCES:
- [Background] Baylor CR, Yorkston KM, Eadie TL. The consequences of spasmodic dysphonia on communication-related quality of life: a qualitative study of the insider's experiences. J Commun Disord. 2005 Sep-Oct;38(5):395-419. doi: 10.1016/j.jcomdis.2005.03.003. PMID 15963338
- [Background] Gaskill CS, Awan JA, Watts CR, Awan SN. Acoustic and Perceptual Classification of Within-sample Normal, Intermittently Dysphonic, and Consistently Dysphonic Voice Types. J Voice. 2017 Mar;31(2):218-228. doi: 10.1016/j.jvoice.2016.04.016. Epub 2016 May 27. PMID 27241579
- [Background] Ludlow CL, Naunton RF, Terada S, Anderson BJ. Successful treatment of selected cases of abductor spasmodic dysphonia using botulinum toxin injection. Otolaryngol Head Neck Surg. 1991 Jun;104(6):849-55. doi: 10.1177/019459989110400614. PMID 1908979
- [Background] Ali SO, Thomassen M, Schulz GM, Hosey LA, Varga M, Ludlow CL, Braun AR. Alterations in CNS activity induced by botulinum toxin treatment in spasmodic dysphonia: an H215O PET study. J Speech Lang Hear Res. 2006 Oct;49(5):1127-46. doi: 10.1044/1092-4388(2006/081). PMID 17077220
- [Background] Norris SA, Morris AE, Campbell MC, Karimi M, Adeyemo B, Paniello RC, Snyder AZ, Petersen SE, Mink JW, Perlmutter JS. Regional, not global, functional connectivity contributes to isolated focal dystonia. Neurology. 2020 Oct 20;95(16):e2246-e2258. doi: 10.1212/WNL.0000000000010791. Epub 2020 Sep 10. PMID 32913023
- [Background] Simonyan K, Ludlow CL. Abnormal activation of the primary somatosensory cortex in spasmodic dysphonia: an fMRI study. Cereb Cortex. 2010 Nov;20(11):2749-59. doi: 10.1093/cercor/bhq023. Epub 2010 Mar 1. PMID 20194686
- [Background] Chen M, Summers RLS, Prudente CN, Goding GS, Samargia-Grivette S, Ludlow CL, Kimberley TJ. Transcranial magnetic stimulation and functional magnet resonance imaging evaluation of adductor spasmodic dysphonia during phonation. Brain Stimul. 2020 May-Jun;13(3):908-915. doi: 10.1016/j.brs.2020.03.003. Epub 2020 Mar 13. PMID 32289724
- [Background] Erickson ML. Effects of voicing and syntactic complexity on sign expression in adductor spasmodic dysphonia. Am J Speech Lang Pathol. 2003 Nov;12(4):416-24. doi: 10.1044/1058-0360(2003/087). PMID 14658993
- [Background] Hirano M, Ohala J. Use of hooked-wire electrodes for electromyography of the intrinsic laryngeal muscles. J Speech Hear Res. 1969 Jun;12(2):362-73. doi: 10.1044/jshr.1202.362. No abstract available. PMID 5808863
- [Background] Chen M, Deng H, Schmidt RL, Kimberley TJ. Low-Frequency Repetitive Transcranial Magnetic Stimulation Targeted to Premotor Cortex Followed by Primary Motor Cortex Modulates Excitability Differently Than Premotor Cortex or Primary Motor Cortex Stimulation Alone. Neuromodulation. 2015 Dec;18(8):678-85. doi: 10.1111/ner.12337. Epub 2015 Aug 26. PMID 26307511
- [Background] Chen M, Summers RL, Goding GS, Samargia S, Ludlow CL, Prudente CN, Kimberley TJ. Evaluation of the Cortical Silent Period of the Laryngeal Motor Cortex in Healthy Individuals. Front Neurosci. 2017 Mar 7;11:88. doi: 10.3389/fnins.2017.00088. eCollection 2017. PMID 28326007
- [Background] Bradnam LV, Stinear CM, Lewis GN, Byblow WD. Task-dependent modulation of inputs to proximal upper limb following transcranial direct current stimulation of primary motor cortex. J Neurophysiol. 2010 May;103(5):2382-9. doi: 10.1152/jn.01046.2009. Epub 2010 Mar 10. PMID 20220073
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Siebner HR, Filipovic SR, Rowe JB, Cordivari C, Gerschlager W, Rothwell JC, Frackowiak RS, Bhatia KP. Patients with focal arm dystonia have increased sensitivity to slow-frequency repetitive TMS of the dorsal premotor cortex. Brain. 2003 Dec;126(Pt 12):2710-25. doi: 10.1093/brain/awg282. Epub 2003 Aug 22. PMID 12937071
- [Background] Murase N, Rothwell JC, Kaji R, Urushihara R, Nakamura K, Murayama N, Igasaki T, Sakata-Igasaki M, Mima T, Ikeda A, Shibasaki H. Subthreshold low-frequency repetitive transcranial magnetic stimulation over the premotor cortex modulates writer's cramp. Brain. 2005 Jan;128(Pt 1):104-15. doi: 10.1093/brain/awh315. Epub 2004 Oct 13. PMID 15483042
- [Background] Lozeron P, Poujois A, Richard A, Masmoudi S, Meppiel E, Woimant F, Kubis N. Contribution of TMS and rTMS in the Understanding of the Pathophysiology and in the Treatment of Dystonia. Front Neural Circuits. 2016 Nov 10;10:90. doi: 10.3389/fncir.2016.00090. eCollection 2016. PMID 27891079
- See also: Link to more information on the study or to contact us. — https://rally.massgeneralbrigham.org/study/rtms